CLINICAL TRIAL: NCT00323791
Title: A Phase II Trial of Gemzar (Gemcitabine) and Gleevec (Imatinib Mesylate) in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Gemcitabine With or Without Imatinib Mesylate in Treating Patients With Metastatic or Unresectable Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Mark Stein, MD, UMDNJ/CINJ
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000539400; P30CA072720 (NIH); CINJ-080507; CINJ-5633; CINJ-NJ3805
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; clear cell renal cell carcinoma; papillary renal cell carcinoma; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Gemcitabine; Imatinib Mesylate; Gene Expression Profiling; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: imatinib mesylate
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine together with imatinib mesylate may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying gemcitabine and imatinib mesylate to see how well they work compared with gemcitabine alone in treating patients with metastatic or unresectable kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare stable disease and objective response in patients with metastatic or unresectable renal cell carcinoma treated with gemcitabine hydrochloride with or without imatinib mesylate.

Secondary

* Evaluate the median survival, progression-free survival, and response rate in patients treated with gemcitabine hydrochloride and imatinib mesylate.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Determine the expression of c-KIT and platelet-derived growth factor receptor-alpha protein expression in both tumor cells and associated endothelial cells using immunohistochemistry staining of paraffin-embedded tissue.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by histology (clear cell vs nonclear cell) and prior therapy (immunotherapy/chemotherapy vs targeted agents).

Patients receive gemcitabine hydrochloride IV on days 3 and 10 and oral imatinib mesylate on days 1-5 and 8-12. Treatment repeats every 21 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving partial or complete response after 2 courses of treatment continue treatment with gemcitabine hydrochloride and imatinib mesylate in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 2 courses of treatment are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV on days 3 and 10.
* Arm II: Patients receive gemcitabine hydrochloride IV on days 3 and 10 and oral imatinib mesylate on days 1-5 and 8-12.

In both arms, treatment repeats every 21 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.

Available archived tumor tissue samples are obtained for immunohistochemical analysis to quantify the expression of c-KIT and platelet-derived growth factor receptor-alpha protein expression.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma

  * Metastatic disease OR unresectable primary tumor
  * No known curative therapy exists
* Documented progressive renal cell carcinoma as defined by RECIST criteria within the past 6 months
* Measurable disease with ≥ 1 unidimensionally measurable lesion
* No known symptomatic brain metastasis or untreated brain metastases or carcinomatous meningitis

  * Treated brain metastasis allowed provided the following criteria are met:

    * Clinically stable
    * More than 7 days since prior steroids

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception during and for 3 months after completion of study treatment
* Must be able to swallow oral medication
* No coexisting medical condition that would preclude study compliance
* No history of allergic reaction to compounds of similar chemical or biological composition to gemcitabine hydrochloride and/or imatinib mesylate
* No uncontrolled illness that would preclude study participation
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia requiring therapy
* No myocardial infarction within the past 6 months
* No active infection
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanoma skin cancer
* No New York Heart Association class III-IV congestive heart failure
* No known chronic liver disease (i.e., chronic active hepatitis or cirrhosis)
* No known HIV positivity
* No significant history of noncompliance to medical regimens

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* No more than 3 prior treatment regimens, including any of the following:

  * No more than 1 prior cytotoxic therapy
  * Immunotherapy regimens comprising interferon and/or aldesleukin
  * Therapy with molecular targets
  * Any combination of the above treatments to a maximum of 3 total therapies
* No prior gemcitabine hydrochloride for metastatic disease
* No prior imatinib mesylate for metastatic disease
* More than 2 weeks since prior major surgery
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 3 weeks since prior anti-vascular endothelial growth factor therapy
* At least 3 weeks since prior radiotherapy

  * Must have evidence of ≥ 1 measurable target lesion outside the radiation fields OR radiologically confirmed disease progression within the radiation fields after completion of radiotherapy
* At least 28 days since prior and no other concurrent investigational or commercial agents, unless disease is rapidly progressing
* No concurrent therapeutic warfarin

  * Concurrent low molecular weight heparin or heparin allowed for therapeutic anticoagulation
  * Concurrent prophylactic warfarin therapy ≤ 1 mg daily to maintain catheter patency allowed
* No concurrent filgrastim (G-CSF) for prevention of neutropenia
* No other concurrent chemotherapy, immunotherapy, hormonal cancer therapy, radiation therapy, or cancer surgery
* No concurrent routine use (i.e., daily or every other day) of systemic corticosteroid therapy (in supraphysiologic doses)
* No concurrent medication that would preclude study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Stable disease
Objective response

SECONDARY OUTCOMES:
Median survival
Progression-free survival
Response rate
Expression of c-KIT and platelet-derived growth factor receptor-alpha protein expression

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stein, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States